CLINICAL TRIAL: NCT07258134
Title: Negative Pressure Wound Therapy Versus Secondary Intention Healing in Stoma Reversal: A Randomized Controlled Trial Evaluating Surgical Site Infection and Wound Outcomes
Brief Title: Compare Stoma Reversal Wound Outcomes Between NPWT and Secondary Intention Healing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sindh Institute of Urology and Transplantation (Other)
Responsible Party: Principal Investigator, Muammad Arsalan Khan, Professor, Sindh Institute of Urology and Transplantation
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SIUT-ERC-2025/A-275
Record Dates: First submitted 2025-09-23; First posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Negative-Pressure Wound Therapy; Wound Heal; Stoma Site Infection; Surgical Site Infection
Keywords: Negative pressure wound therapy; secondary intention Healing; Surgical site infection; asepsis score
MeSH Terms: conditions — Surgical Wound Infection | interventions — Negative-Pressure Wound Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Negative pressure wound therapy (Experimental): In the NPWT (negative-pressure wound therapy) group, after the procedure, the skin was left open and covered with four sterile gauze layers. An 18 Fr Nelaton catheter was placed directly over the wound and sealed with transparent, waterproof adhesive to create a vacuum. Continuous negative pressure was applied at 15 mmHg. Dressings were evaluated for Surgical site infection on postoperative days 2 and 4 using the ASEPSIS score; if no infection was present, a NPWT dressing was reapplied. On postoperative day 6, a final wound assessment was conducted, and further management was carried out as per departmental protocol.
  Interventions: Procedure: Negative Pressure Wound Therapy
- secondary intention healing (No Intervention): In the SIH (secondary intention healing) group, the wound was left open and dressed using four layers of sterile gauze and a transparent adhesive dressing. Similar to the NPWT group, dressing changes and assessments using the ASEPSIS score were performed on postoperative days 2, 4, and 6. If an infection was identified, standard management protocols were followed.

INTERVENTIONS:
Procedure: Negative Pressure Wound Therapy — In the NPWT (negative pressure wound therapy) group, after the procedure, the skin was left open and covered with four sterile gauze layers. An 18 Fr Nelaton catheter was placed directly over the wound and sealed with transparent, waterproof adhesive to create a vacuum. Continuous negative pressure was applied at 15 mmHg. Dressings were evaluated for SSI on postoperative days 2 and 4 using the ASEPSIS score; if no infection was present, NPWT dressing was reapplied. On postoperative day 6, final wound assessment was conducted and further management was carried out as per departmental protocol.
  Arms: Negative pressure wound therapy

SUMMARY:
This was a single-center, parallel-group randomized controlled trial conducted in 2024 at the General Surgery Ward of the Sindh Institute of Urology and Transplantation (SIUT), Karachi. The study compared negative pressure wound therapy (NPWT) with healing by secondary intention (SIH) for patients undergoing stoma reversal surgery.

DETAILED DESCRIPTION:
Study Design and Participants A total of 92 adult patients (aged ≥18 years) scheduled for stoma reversal were assessed for eligibility. Of these, 72 patients who met the inclusion criteria and provided informed consent were enrolled and randomized in a 1:1 ratio into NPWT (intervention) and SIH (control) groups (n=36 each). Eligibility criteria included patients undergoing elective or emergency stoma reversal with conventional layered closure of the muscular layer and skin management by either NPWT or SIH. Exclusion criteria included use of skin closure techniques other than suture, prolonged antibiotic use before surgery, or need for reoperation for causes other than surgical site infection (SSI).

Randomization and Allocation Random allocation was performed using simple random sampling by lot draw. A list of consecutive serial numbers with equal halves of even and odd numbers was utilized. Each number was printed separately on slips of paper and folded to conceal. A slip was drawn for each patients allocation. Patients who drew odd-numbered lots were assigned to the treatment group (NPWT), and those with even-numbered lots to the control group (SIH). This approach ensured unbiased allocation while maintaining transparency.

Interventions In both groups, stoma reversal was performed following standard operative protocols with fascial layer closure using absorbable sutures. In the NPWT group, after the procedure, the skin was left open and covered with four sterile gauze layers. An 18 Fr Nelaton catheter was placed directly over the wound and sealed with transparent, waterproof adhesive to create a vacuum. Continuous negative pressure was applied at 15 mmHg. Dressings were evaluated for SSI on postoperative days 2 and 4 using the ASEPSIS score; if no infection was present, the NPWT dressing was reapplied. On postoperative day 6, a final wound assessment was conducted, and further management was carried out as per departmental protocol.

In the SIH group, the wound was left open and dressed using four layers of sterile gauze and a transparent adhesive dressing. Similar to the NPWT group, dressing changes and assessments using the ASEPSIS score were performed on postoperative days 2, 4, and 6. If an infection was identified, standard management protocols were followed.

All patients received prophylactic antibiotics with piperacillin-tazobactam (4.5 g) administered 30 minutes before incision and three postoperative doses of the same antibiotic.

ELIGIBILITY:
Inclusion Criteria:

All patients aged between 18-80 years undergoing stoma reversal surgery were included, following their formal consent for inclusion in the study protocol.

Exclusion Criteria:

* Patients with history of prolonged antibiotic use prior to stoma reversal surgery (>1months).
* Patients with prior skin condition that required medical treatment (for instance, Plaque Psoriasis).
* Patient with prior history of wound-related complication (like keloids or hypertrophic scars).

Furthermore, after allocation, the patients with the following protocol violations were also excluded:

* Patients who had undergone any other forms of wound closure after stoma reversal, that deviated from the study protocol.
* Patients who were re-operated during the hospital stay for any other reason than surgical site infection.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2025-02-24 (Actual); Primary Completion 2025-08-30 (Actual); Study Completion 2025-08-30 (Actual)

PRIMARY OUTCOMES:
Highest Postoperative Asepsis Score for SSI assessment | Post-operative day (POD) 2, 4 and 6 (ASEPSIS score recorded)
  The primary outcome was the occurrence and severity of surgical site infection, assessed using the ASEPSIS scoring system (Additional treatment, Serous discharge, Erythema, Purulent exudate, Separation of deep tissues, Isolation of bacteria, and Stay duration as an inpatient) on postoperative days 2, 4, and 6. The highest ASEPSIS score recorded across these time points was used for between-group comparison. The score may vary between. 0-70 with higher score representing worse outcome.

SECONDARY OUTCOMES:
Scar Cosmesis Assessment and Rating (SCAR) score on postoperative day 30 | On Postoperative day 30 wound cosmesis were assessed using scar scale
  All patient's operative wounds were assessed for cosmesis on postoperative day 30. This was performed utilizing the Scar Cosmesis Assessment and Rating (SCAR) scale for objective assessment. Scores range from 0 (best possible scar) to 15 (worst possible scar).
Length of Stay | 6-12 days. Following completion of study observations on postoperative day 6, patient may be discharged on meeting the discharge criteria. Expected between 6-12 days.
  Duration of stay assessed as: number of days of hospital stay after the index procedure till the patient discharged from hospital was recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Sindh Institute of Urology and Transplantation, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided